CLINICAL TRIAL: NCT01634594
Title: The Effect of Deliberate Hypotension on QTc, Tp-e Intervals and Heart Rate Variability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2012-0242
Record Dates: First submitted 2012-06-25; First posted 2012-07-06 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Mandibular Prognathism; Mandibular Retrognathism
Keywords: Deliberate hypotension, QTc, Tp-e, heart rate variability
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- sevoflurane-remifentanil (group R) (Experimental): Continuous infusion of remifentanil at 0.05 ~ 2 mcg/kg/min with sevoflurane concentration of 1 MAC
  Interventions: Drug: Group R
- sevoflurane-nicardipine (group N) (Active Comparator): Continuous infusion of nicardipine at 1 ~ 7 mcg/kg/min with sevoflurane concentration of 1 MAC
  Interventions: Drug: Group N
- sevoflurane-dexmedetomidine (group D) (Active Comparator): Continuous infusion of dexmedetomidine at 0.2 ~ 1.0 mcg/kg/hr with sevoflurane concentration of 1 MAC
  Interventions: Drug: Group D

INTERVENTIONS:
Drug: Group R
  Other Names: Continuous infusion of remifentanil at 0.05 ~ 2 mcg/kg/min with sevoflurane concentration of 1 MAC
  Arms: sevoflurane-remifentanil (group R)
Drug: Group N
  Other Names: Continuous infusion of nicardipine at 1 ~ 7 mcg/kg/min with sevoflurane concentration of 1 MAC
  Arms: sevoflurane-nicardipine (group N)
Drug: Group D
  Other Names: Continuous infustion of dexmedetomidine at 0.2 ~ 1.0 mcg/kg/hr with sevoflurane concentration of 1 MAC
  Arms: sevoflurane-dexmedetomidine (group D)

SUMMARY:
Deliberate hypotension is defined as lowering the systolic blood pressure to 80-90mmHg, or the mean blood pressure to 50-65mmHg. This technique is usually employed for operations that have a high risk of intraoperative hemorrhage, such as orthognathic surgery. Several different regimens are used to lower the patient's blood pressure, such as vasodilators, autonomic nervous system inhibitors, opioids and inhalation anesthetics. However, the effects that these agents have on the QTc and Tp-e intervals during deliberate hypotension is not known. Virtually every kind of anesthetic is reported to have some effect on the QTc and Tp-e intervals. Because orthognathic surgery usually takes 3-4 hours to complete, the amount of anesthetics and drugs used to maintain low blood pressure is not small. Therefore, the effect that these agents may have on the QTc and Tp-e intervals may not be negligible. The investigators of the present study found that the high dose of commonly used hypotensive agents tend to prolong these variabilities to some extent. This study will be able to provide insight as to which hypotensive anesthesia regimen has the least effect on the QTc and Tp-e intervals, and therefore will be helpful in minimizing cardiovascular risks of deliberate hypotensive anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class 1
2. Adults over the age of 20
3. Patients requiring deliberate hypotensive anesthesia for orthognathic surgery

Exclusion Criteria:

1. Patient refusal
2. Patients with arrhythmia
3. Patients with cardiac anomalies or past history of cardiac surgery
4. Patients with abnormal electrolyte levels
5. Patients taking medications that are known to prolong QT intervals
6. Patients with QTc intervals greater than 440ms
7. Illiterate patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Changes in QTc, Tp-e interval during deliberate hypotension | Before induction of anesthesia (T1), 10 minutes after induction of anesthesia (T2), 30 minutes after target blood pressure is reached (T3), every 60 minutes after from the end of surgery

SECONDARY OUTCOMES:
Changes in Tp-e interval during deliberate hypotension | Before induction of anesthesia (T1), 10 minutes after induction of anesthesia (T2), 30 minutes after target blood pressure is reached (T3), every 60 minutes after from the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Young Jun Oh, Seoul, South Korea